CLINICAL TRIAL: NCT04705415
Title: A Randomized, Double-Blind, Single and Multiple Ascending Dose Study to Assess the Safety and Pharmacokinetics of Niclosamide in Healthy Adults
Brief Title: A Single and Multiple Ascending Dose Study of Niclosamide in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroBo Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ANA001-002
Record Dates: First submitted 2020-12-08; First posted 2021-01-12 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Niclosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomized, Double-Blind Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- SAD Cohort 1: ANA001 1000 mg po (Experimental): Subjects will receive a 1000 mg single oral dose of ANA001 with a standardized light meal presented at 4 x 250 mg capsules. Each capsule is 250 mg.
  Interventions: Drug: Niclosamide
- SAD Cohort 2: ANA001 2000 mg po (Experimental): Subjects will a 2000 mg single oral dose of ANA001 with a standardized light meal presented at 8 x 250 mg capsules. Each capsule is 250 mg.
  Interventions: Drug: Niclosamide
- SAD Cohort 3: ANA001 3000 mg po (Experimental): Subjects will a 3000 mg single oral dose of ANA001 with a standardized light meal presented at 12 x 250 mg capsules. Each capsule is 250 mg.
  Interventions: Drug: Niclosamide
- SAD Cohorts 1, 2 & 3: Pooled Matching Placebo (Placebo Comparator): Subjects will receive matching placebo hydroxypropylmethylcellulose (HPMC) as a single oral dose (4, 8, or 12 capsules) with a standardized light meal.
  Interventions: Drug: Placebo
- MAD Cohort 1: ANA001 1000 mg po BID (Experimental): Subjects will receive an oral dose of 1000mg ANA001 twice daily (BID) with a standardized light meal for 7 consecutive days. Each dose will be presented as 4 250mg capsules.
  Interventions: Drug: Niclosamide
- MAD Cohort 2: ANA001 1000 mg po TID (Experimental): Subjects will receive an oral dose of 1000mg ANA001 three times daily (TID) with a standardized light meal for 7 consecutive days. Each dose will be presented as 4 250mg capsules.
  Interventions: Drug: Niclosamide
- MAD Cohorts 1 & 2: Pooled Matching Placebo (Placebo Comparator): Subjects will receive an oral dose of matching Placebo to ANA001 two (BID) three times daily (TID) with a standardized light meal for 7 consecutive days. Each dose will be presented as 4 250mg capsules of hydroxypropylmethylcellulose (HPMC)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Niclosamide — Niclosamide is an antihelmintic with in-vitro antiviral activity
  Other Names: ANA001
  Arms: MAD Cohort 1: ANA001 1000 mg po BID; MAD Cohort 2: ANA001 1000 mg po TID; SAD Cohort 1: ANA001 1000 mg po; SAD Cohort 2: ANA001 2000 mg po; SAD Cohort 3: ANA001 3000 mg po
Drug: Placebo — Matching hydroxypropylmethylcellulose HPMC capsules with no active ingredients
  Other Names: Matching Placebo to ANA001
  Arms: MAD Cohorts 1 & 2: Pooled Matching Placebo; SAD Cohorts 1, 2 & 3: Pooled Matching Placebo

SUMMARY:
A single and multiple ascending dose study of ANA001 in healthy adults to assess the safety and pharmacokinetics

DETAILED DESCRIPTION:
This is a Phase 1, single center, randomized, double blind, single ascending dose (SAD) and multiple ascending dose (MAD) study to assess the safety and pharmacokinetics of ANA001 in healthy adult subjects. In the single ascending dose portion of the study, subjects in 3 cohorts of 10 subjects each will be randomized to receive a single daily oral dose of ANA001 or matching placebo. In the multiple ascending dose portion of the study, subjects in 3 cohorts of 12 subjects each will be randomized to receive twice or thrice daily oral dose of ANA001 or matching placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the study informed consent form
2. Man or woman, 18 to 65 years of age inclusive at the time of signing the informed consent form
3. Overtly healthy as determined by medical evaluation
4. Body mass index (BMI) within 18 to 30.0 kg/m2 (inclusive) and body weight not less than 50 kg
5. Blood pressure at Screening and Day -1 between 90 and 140 mmHg systolic, inclusive, and no higher than 90 mmHg diastolic.
6. A 12-lead electrocardiogram (ECG) at Screening consistent with normal cardiac conduction and function, including:

   * Sinus rhythm
   * Pulse rate between 50 and 100 beats per minute (bpm)
   * QTc interval 450 milliseconds (QT interval corrected using Fridericia correction method [QTcF])
   * QRS interval of <120 milliseconds
   * PR interval <200 milliseconds
   * Morphology consistent with healthy cardiac conduction and function
7. Non-smoker or ex-smoker for >12 months
8. If male, must agree to use contraception methods outlined for the study during the treatment period and for at least 30 days (a spermatogenesis cycle) after the last dose of study treatment and refrain from donating sperm during this period
9. If female, is not pregnant, not breastfeeding, and meets at least one of the following conditions:

Not a woman of childbearing potential (WOCBP)

OR

A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 30 days (one menstrual cycle) after the last dose of study treatment.

Exclusion Criteria:

1. Has a history of or current clinically significant medical illness including but not limited to, cardiac arrhythmias or other cardiac disease; hematologic disease; coagulation disorders (including any abnormal bleeding or blood dyscrasias); lipid abnormalities; significant pulmonary disease, including bronchospastic respiratory disease; diabetes mellitus; hepatic or renal insufficiency (creatinine clearance below 60 mL/min); thyroid disease; neurologic or psychiatric disease; infection; or any other illness that the Investigator considers should exclude the subject or that could interfere with the interpretation of the study results.
2. Has known allergy to niclosamide or salicylate-containing medications.
3. Clinically significant abnormal values for hematology, clinical chemistry, or urinalysis at screening.
4. Clinically significant abnormal physical examination, vital signs or 12 lead ECG at screening.
5. Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV; has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening.
6. History of drug or alcohol abuse according to Diagnostic and Statistical Manual of Mental Disorders (4th edition) criteria within 5 years before screening or positive test result(s) for alcohol and/or drugs of abuse at screening and admission
7. Has received an investigational drug or used an invasive investigational medical device within 1 month or within a period less than 10 times the drug's half-life, whichever is longer, before Day 1.
8. Has preplanned surgery or procedures that would interfere with the conduct of the study
9. Is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, as well as family members of the employees or the Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Doug Rank, MD, Study Director — NeuroBo Pharmaceuticals Inc.
Locations (1):
- WCCT Global Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- SAD Cohorts 1, 2 & 3: Pooled Matching Placebo: For the single ascending dose (SAD) portion of the study, subjects will receive matching placebo hydroxypropylmethylcellulose (HPMC) as a single oral dose (4, 8, or 12 capsules) with a standardized light meal.
  Placebo: Matching hydroxypropylmethylcellulose HPMC capsules with no active ingredients
Period: Overall Study
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Started | 8 | 8 | 8 | 6 | 9 | 9 | 6
Completed | 7 | 7 | 8 | 5 | 8 | 9 | 5
Not Completed | 1 | 1 | 0 | 1 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- SAD Cohorts 1, 2 & 3: Pooled Matching Placebo: A matching placebo to a single oral 3000mg dose of 1000mg was administered with a standardized light meal (500 to 750 cal) after an overnight fast of at least 10 hours.
- Total: Total of all reporting groups
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo | Total
Number analyzed (Participants) | 8 | 8 | 8 | 6 | 9 | 9 | 6 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 6 | 9 | 9 | 6 | 54
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (13.9) | 41.6 (16.3) | 45.8 (11.6) | 47.2 (12.8) | 45.8 (13.3) | 41.8 (12.4) | 38.2 (6) | 43.6 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 4 | 3 | 5 | 4 | 3 | 24
  Male | 7 | 4 | 4 | 3 | 4 | 5 | 3 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 2 | 1 | 3 | 2 | 1 | 16
  Not Hispanic or Latino | 5 | 4 | 6 | 5 | 6 | 7 | 5 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 0 | 3 | 3 | 3 | 11
  White | 5 | 6 | 6 | 3 | 6 | 5 | 1 | 32
  More than one race | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 6 | 9 | 9 | 6 | 54

OUTCOME MEASURES:

1. Primary Outcome: SAD: Number of Subjects Reporting TEAEs and STEAEs
Description: Number of Subjects Reporting treatment-emergent AEs (TEAEs) and Serious treatment-emergent AEs (STEAEs) in the SAD
Time Frame: Baseline to Day 7.
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants
  Number of Subjects Reporting treatment-emergent AEs (TEAEs) | 0 | 0 | 0 | 1
  Number of Subjects Reporting treatment-emergent Serious AEs (STEAEs) | 0 | 0 | 0 | 0

2. Primary Outcome: MAD: Number of Subjects Reporting TEAEs and STEAEs
Description: Number of Subjects Reporting treatment-emergent AEs (TEAEs) and Serious treatment-emergent AEs (STEAEs) in the MAD
Time Frame: Baseline to Day 14.
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants
  Number of Subjects Reporting TEAEs | 3 | 3 | 1
  Number of Subjects Reporting STEAEs | 0 | 0 | 0

3. Primary Outcome: SAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in ECG Parameters
Description: Number of Subjects with Clinically Significant changes in ECG parameters from Baseline (PR, QRS, QT, and QTc intervals)
Time Frame: Baseline to Day 7
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0

4. Primary Outcome: MAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in ECG Parameters
Description: Number of Subjects with Clinically Significant changes in ECG parameters from Baseline (PR, QRS, QT, and QTc intervals)
Time Frame: Baseline to Day 14
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants | 0 | 0 | 0

5. Primary Outcome: SAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Haematology
Description: Number of Subjects with Clinically Significant changes in Haematology (Basophils (%),Eosinophils (%, Ery. Mean Corpuscular Hemoglobin, Ery. Mean Corpuscular Volume, Erythrocytes (10^12/L), Hematocrit (%), Hemoglobin (g/dL). Hemoglobin (g/dL), Lymphocytes (%), Monocytes (%), Neutrophils (%)' Platelets (10^9/L), Reticulocytes (%))
Time Frame: Baseline to Day 7
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0

6. Primary Outcome: MAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Haematology
Description: as for outcome 5
Time Frame: Baseline to Day 14
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants | 0 | 0 | 0

7. Primary Outcome: SAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Serum Chemistry
Description: Number of Subjects with Clinically Significant changes in Serum Chemistry (Alanine Aminotransferase (U/L), Alkaline Phosphatase (U/L), Aspartate Aminotransferase (U/L), Bilirubin (mg/dL), Calcium (mg/dL), Creatinine (mg/dL), Direct Bilirubin (mg/dL, Glucose (mg/dL), Potassium (mmol/L), Protein (g/dL), Sodium (mmol/L), Urea Nitrogen (mg/dL)
Time Frame: Baseline to Day 7
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0

8. Primary Outcome: MAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Serum Chemistry
Description: as for outcome 7
Time Frame: Baseline to Day 14
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants | 0 | 0 | 0

9. Primary Outcome: SAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Urinalysis
Description: Number of Subjects with Clinically Significant changes in Urinalysis (Specific Gravity, Urobilinogen (EU), pH)
Time Frame: Baseline to Day 7
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0

10. Primary Outcome: MAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Urinalysis
Description: Number of Subjects with Clinically Significant changes in Urinalysis (Specific Gravity, Urobilinogen (EU), pH)
Time Frame: Baseline to Day 14
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants | 0 | 0 | 0

11. Primary Outcome: SAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Vital Signs
Description: Number of Subjects with Clinically Significant changes in Vital Signs from Baseline (Diastolic Blood Pressure, Systolic Blood Pressure (mmHg), Pulse Rate (beats/min), Respiratory Rate (breaths/min))
Time Frame: Baseline to Day 7
Measure: Number; unit: participants
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 6
participants | 0 | 0 | 0 | 0

12. Primary Outcome: MAD: Safety and Tolerability of ANA001 as Measured by Clinically Significant Changes in Vital Signs
Description: as for outcome 11
Time Frame: Baseline to Day 14
Measure: Number; unit: participants
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
Number analyzed (Participants) | 9 | 9 | 6
participants | 0 | 0 | 0

13. Secondary Outcome: SAD: Tmax
Description: Time to reach the maximum plasma concentration (SAD)
Time Frame: PK samples were collected before dosing and at 0.5, 1, 2, 4, 6, 8, 10, 12 and 24 hours. A Follow-up sample was taken Day 7 (±2) after dosing.
Measure: Median (Full Range); unit: h
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
h | 4 [4 to 8] | 4 [4 to 10] | 4 [2 to 4.02]

14. Secondary Outcome: SAD: Cmax
Description: Maximum plasma concentration during a dosing interval (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
ng/mL | 328 (230) | 647 (306) | 347 (124)

15. Secondary Outcome: SAD: AUC0-t
Description: Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentration (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 1420 (889) | 4620 (2040) | 1780 (558)

16. Secondary Outcome: SAD: AUC0-∞
Description: Area under the plasma concentration time curve from time 0 extrapolated to infinity, calculated as AUC0-last + Clast/λ, where Clast is the last quantifiable concentration at time t (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
h*ng/mL | 1660 (985) | 4890 (2310) | 1860 (575)

17. Secondary Outcome: SAD: t1/2
Description: Elimination half-life associated with the terminal slope (λ) of the semilogarithmic drug concentration-time curve, calculated as 0.693/λ (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
h | 4.40 (2.30) | 3.30 (0.925) | 5.34 (2.24)

18. Secondary Outcome: SAD: CL/F
Description: Systemic Clearance (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
L/h | 940 (631) | 572 (397) | 1780 (705)

19. Secondary Outcome: SAD: Vz/F
Description: Volume of distribution (SAD)
Time Frame: as for outcome 13
Measure: Mean (Standard Deviation); unit: L
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po
Number analyzed (Participants) | 8 | 8 | 8
L | 8540 (9010) | 3210 (3190) | 15100 (9390)

20. Secondary Outcome: MAD: Tmax Day 1
Description: Time to reach the maximum plasma concentration Day 1
Time Frame: BID: Samples on Days 1 and 7 before dosing and at 0.5, 1, 2, 4, 6, 8, 10, and 12 hours after dosing; Days 2, 4, 6, and 8 before dosing and before the 12 h. dose on Days 2, 4, and 6.TID: As BID but omitting samples at 10, and 12 hours after dosing.
Measure: Median (Full Range); unit: h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 9
h | 4 [2 to 6.05] | 4 [2 to 6]

21. Secondary Outcome: MAD: Tmax Day 7
Description: Time to reach the maximum plasma concentration (Day 7)
Time Frame: as for outcome 20
Measure: Median (Full Range); unit: h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 9
h | 4 [2 to 6] | 2 [2 to 6]

22. Secondary Outcome: MAD: Cmax Day 1
Description: Maximum plasma concentration during a dosing interval (Day 1)
Time Frame: BID: Samples on Days 1 and 7 before dosing and at 0.5, 1, 2, 4, 6, 8, 10, and 12 hours after dosing; Days 2, 4, 6, and 8 before dosing and before the 12 h. dose on Days 2, 4, and 6.TID: For BID but omitting samples at 10, and 12 hours after dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 8
ng/mL | 332 (110) | 259 (158)

23. Secondary Outcome: MAD: Cmax Day 7
Description: Maximum plasma concentration during a dosing interval (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 9
ng/mL | 234 (77.9) | 235 (70.9)

24. Secondary Outcome: MAD: AUC0-t Day 1
Description: Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentration (Day 1)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 9
h*ng/mL | 1630 (499) | 1360 (968)

25. Secondary Outcome: MAD: AUC0-t Day 7
Description: Area under the plasma concentration-time curve from time 0 to time the last quantifiable concentration (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 9
h*ng/mL | 1100 (481) | 993 (250)

26. Secondary Outcome: MAD: AUC0-tau Day 1
Description: Area under the plasma concentration-time curve over the dosing interval at steady-state, calculated from the dosing interval (Day 1)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 9
h*ng/mL | 1630 (500) | 1680 (1810)

27. Secondary Outcome: MAD: AUC0-tau Day 7
Description: Area under the plasma concentration-time curve over the dosing interval at steady-state, calculated from the dosing interval (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 9
h*ng/mL | 1100 (480) | 992 (250)

28. Secondary Outcome: MAD: t1/2 Day 1
Description: Elimination half-life associated with the terminal slope (λ) of the semilogarithmic drug concentration-time curve, calculated as 0.693/λ (Day 1)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 7 | 3
h | 1.8 (0.595) | 4.82 (2.94)

29. Secondary Outcome: MAD: t1/2 Day 7
Description: Elimination half-life associated with the terminal slope (λ) of the semilogarithmic drug concentration-time curve, calculated as 0.693/λ (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 7 | 6
h | 2.83 (1.33) | 2.16 (0.194)

30. Secondary Outcome: MAD: CLss Day 1
Description: Systemic Clearance at steady state (Day 1)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 3
L/h | 677 (246) | 1200 (928)

31. Secondary Outcome: MAD: CLss Day 7
Description: Systemic Clearance at steady state (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 9
L/h | 1060 (410) | 1070 (287)

32. Secondary Outcome: MAD: Vdss Day 1
Description: Volume of distribution at steady state (Day 1)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 9 | 3
L | 1920 (788) | 6200 (3750)

33. Secondary Outcome: MAD: Vdss Day 7
Description: Volume of distribution at steady state (Day 7)
Time Frame: as for outcome 20
Measure: Mean (Standard Deviation); unit: L
Arm/Group | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID
Number analyzed (Participants) | 8 | 7
L | 4080 (2010) | 3590 (874)

ADVERSE EVENTS:
Time Frame: SAD: Adverse Event Collected from Dosing to 7 days after dosing (8 days). MAD: Adverse Event Collected from Dosing on Day 1 to 7 days after final dosing day (15 days).
Arm/Group | SAD Cohort 1: ANA001 1000 mg po | SAD Cohort 2: ANA001 2000 mg po | SAD Cohort 3: ANA001 3000 mg po | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo | MAD Cohort 1: ANA001 1000 mg po BID | MAD Cohort 2: ANA001 1000 mg po TID | MAD Cohorts 1 & 2: Pooled Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/9 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/6 | 0/9 | 0/9 | 0/6
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 1/6 | 3/9 | 3/9 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAD Cohort 1: ANA001 1000 mg po (N=8) | SAD Cohort 2: ANA001 2000 mg po (N=8) | SAD Cohort 3: ANA001 3000 mg po (N=8) | SAD Cohorts 1, 2 & 3: Pooled Matching Placebo (N=6) | MAD Cohort 1: ANA001 1000 mg po BID (N=9) | MAD Cohort 2: ANA001 1000 mg po TID (N=9) | MAD Cohorts 1 & 2: Pooled Matching Placebo (N=6)
Dizziness (Nervous system disorders) | NA | NA | NA | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | NA | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Falling Hair
Rash maculo-papular (Skin and subcutaneous tissue disorders) | NA | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headaches NEC (Nervous system disorders) | NA | NA | NA | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Headache
Abdominal Pain (Gastrointestinal disorders) | NA | NA | NA | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Abdominal Cramps
Haemorrhoids (Gastrointestinal disorders) | NA | NA | NA | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | NA | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Skin Tear
Acne (Respiratory, thoracic and mediastinal disorders) | NA | NA | NA | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Pimples

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-01-09): https://cdn.clinicaltrials.gov/large-docs/15/NCT04705415/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-22): https://cdn.clinicaltrials.gov/large-docs/15/NCT04705415/SAP_001.pdf